CLINICAL TRIAL: NCT05460156
Title: The Bridges Self-management Programme for People With Neuromuscular Diseases: A Hybrid II Effectiveness-implementation Feasibility Study
Brief Title: The Bridges Self-management Programme for People With Neuromuscular Diseases
Acronym: ADAPT-NMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Gita Ramdharry, Principle Investigator, University College London Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 137025
Record Dates: First submitted 2021-04-27; First posted 2022-07-15 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NM Bridges (Experimental): Receive NM Bridges supportive care from trained personnel
  Interventions: Behavioral: Bridges Self-management Support

INTERVENTIONS:
Behavioral: Bridges Self-management Support — Self-management support intervention tailored for people with neuromuscular diseases

SUMMARY:
Objectives:

* To evaluate the feasibility of delivering the Neuromuscular Bridges Self-Management Programme (NM Bridges) in addition to usual care.
* To evaluate the feasibility of an implementation strategy package and identify barriers and facilitators to implementation of NM Bridges at a specialist neuromuscular centre.

Type of trial: A hybrid II feasibility trial Trial design and methods:A hybrid trial which simultaneously investigates both the feasibility of NM Bridges, and the feasibility of a package of implementation strategies.

Trial duration per participant: 4 months Estimated total trial duration: 1 year Planned trial sites: Single site Total number of participants planned: 60 Main inclusion/exclusion criteria: Participants will be over the age of 18, with a diagnosis of neuromuscular disease from a neurologist at the Queen Square Centre for Neuromuscular Diseases (CNMD). Participants will be deemed by healthcare professionals to have the capacity to give informed consent to participate in the research.

Statistical methodology and analysis:

This is a single-arm cohort study of feasibility of the NM Bridges intervention. The primary analysis will be of feasibility of conducting a trial of the intervention within a single pilot site. Secondary analysis will be calculation of effect sizes of patient reported outcome measures (PROMS). The investigators will also be interviewing participants and qualitative analysis methods will be used.

DETAILED DESCRIPTION:
Objectives

1. To explore the feasibility of delivering and evaluating NM Bridges through a single, specialist service:

   1. Feasibility of evaluation

      * To examine the acceptability and performance of candidate outcome measures that consider the priorities, needs, skills and goals of individuals living with NMD to gain data for a future, larger trial. As this is feasibility work, this trial is not powered for efficacy.
      * Explore participant recruitment and retention. (Measured through administrative data and assessment of completeness and quality of the collected data
   2. feasibility of delivery of the NM Bridges intervention

      * Explore acceptability of NM Bridges (to clinicians and participants) when delivered in one-off interactions, as this will be necessary in this new clinical setting, has not been explored in previous trials, and will be required for roll-out to other services. (Explored through semi-structured qualitative interviews).
      * Explore demand for NM Bridges within the service. Explored through semi-structured qualitative interviews)
2. To evaluate the feasibility of an implementation strategy 'package' to implement NM Bridges at a specialist neuromuscular centre • Monitor fidelity of the implementation process (e.g., training, supervision, and informatics)

   * Monitor fidelity to the intervention itself (intervention fidelity) e.g. adherence to the intended program content, and responsiveness, quality and competence in delivering the program.
   * Explore acceptability of the implementation strategy package to clinicians at the specialist centre (Explored through semi-structured qualitative interviews).
   * Identify barriers and facilitators to the implementation strategy package
   * Explore appropriateness and practicability of the implementation strategy package to the specialist clinical service (Explored through semi-structured qualitative interviews).
   * Monitor effect of implementation strategy package on adoption of the intervention
   * Assess the level of system change required needed to integrate the intervention into the existing infrastructure, to help determine whether intervention delivery in this setting is truly feasible. (Explored through semi-structured qualitative interviews).

     3 Trial design This hybrid study will involve testing the feasibility of a clinical intervention (NM Bridges) and a simultaneous testing of the feasibility of an implementation strategy package (informed by NPT), with a view to increasing speed of translation (41). Below, the rationale for our design choices are summarised.

Mixed methods An embedded experimental mixed methods design will be used to address the research questions, and is an often used design when evaluating health services research. An embedded design, where one data set provides a supportive secondary role to the other, is frequently used when researchers need to include a qualitative component within a quantitative study. A sequential two-phase approach will be employed, where the use of qualitative methods post intervention will enable the team to follow up on the participants' experiences of the intervention, and the experiences of staff delivering the intervention.

Outcome measures (Quantitative methods) Outcome measures will be completed at baseline, directly after receiving the intervention and 3 months afterwards. There will be the option for outcome measures to be completed remotely, for participant convenience, and to reduce risk associated with the current COVID-19 pandemic.

Semi-structured interviews (Qualitative methods) Ten participants will be recruited for semi-structured interviews to explore their experiences of receiving NM Bridges. Interviews will be audio recorded and transcribed by an external service, who are approved by UCL for such work (Fingertips Typing Services). Thematic analysis and validation will be undertaken by the PhD student.

Six Queen Square Centre For Neuromuscular Diseases (CNMD) staff will be interviewed at the end of the intervention phase of the study to investigate determinants of implementation behaviour and explore experiences of delivering NM Bridges as part of the clinical service. Themes will include benefits, challenges, suggestions for streamlining delivery, translation to other areas and environments. Interviews will be audio recorded and transcribed by an external service, who are approved by UCL for such work (Fingertips Typing Services). Thematic analysis and validation will be undertaken by the PhD student.

Setting The Queen Square Centre for Neuromuscular Diseases (CNMD) is a specialist research and clinical centre which specifically focuses on genetic and acquired neuromuscular diseases. It provides comprehensive NHS clinical services for over 5,000 patients per year which include a range of specialist neuromuscular clinics and nationally commissioned services.

Participant selection Considering the rare nature of many NMDs, recruitment of a heterogeneous sample for this work could be considered as pragmatic, and may augment the ecological validity of the trial, as this is what the day-to-day clinics in a specialist NMD centre are realistically likely to look like.

Staff Training The training for 6 members of the CNMD clinical team has been costed into this grant, and as such, 6 health professionals from the centre will receive Bridges Self-Management training. An education training package specific to the clinical and organisational context has been co-produced with key stakeholders (patients, occupational therapists, physiotherapists and specialist nurses at the CNMD), in order to ensure the training is reflective, sensitive and tailored to the unique environment in which it will be delivered.

Delivery The intervention will be delivered in a one-off session as part of routine therapy and nursing appointments. The intervention is designed to be woven into routine clinical appointments, it is therefore not expected that delivering NM Bridges will have any adverse effect on the time it takes to deliver appointments, the care that participants receive, or the workload of clinicians.

Patient recruitment at a site will only commence once evidence of the following approval/essential documents are in place:

Participant recruitment at a site will only commence when the trial has:

1. Been confirmed by the Sponsor (or it's delegated representative), and
2. Been issued an 'NHS permission letter'.
3. Has regulatory body approval from REC and HRA.

Patients with NMD attending the CNMD clinics will be invited to participate by the PI or other members of the clinical care team. The PI is part of the clinical care team. Suitable patients will be approached by the clinical care team or research team during routine clinics. The initial approach will only be done by a member of the clinical team. The purpose of the study will be explained, the terms of participation and any queries answered. A PIS (reviewed by a PPI group set up specifically for the study) will be handed out to all those interested in the study. The research team will follow up interested patients wishing to consider their participation. Permission will be sought to contact interested patients, contact details will be taken and they will be sent a study information sheet to review in their own time. Participants may also be recruited from physiotherapy clinics at the National Hospital for Neurology and Neurosurgery.

The clinical care team will identify potential participants who will be sent a letter of invitation to participate, a study information sheet and details of how to register interest in the study by telephone, email or letter. On receipt of an expression of interest, contact will be made with the patient by a member of the research team.

Interested patients will be given at least one week to consider the study before they are asked to decide whether to take part.

4 Informed consent A copy of the signed Informed Consent form will be given to the participant. The original signed form will be retained in the trial file at site and a copy placed in the medical notes. This will also be the case for remote consent.

Product/Interventions

1. Name and description of intervention under investigation

   Neuromuscular Bridges Self-Management Support Programme (NM Bridges) NM Bridges is a co-produced intervention delivered to individual service users by healthcare professionals, and supported by a patient held workbook. NM Bridges is an adaptation adapted of the original programme for individuals with stroke. It is based on the principle of self-efficacy, defined as ''the belief in one's capabilities to organize and execute the courses of action required to produce given attainments''. More information on the history and development of Bridges is found in the background section under NM Bridges

   Overview of the Bridges self-management package:

   Training for practitioners including:

   • Theory, research and practical examples relating to stroke and self-management
   * Debate and discussion about integration into practice, using case-based examples
   * Practice using Bridges principles and patient workbook
   * Completion of case reflections from using NM Bridges in practice
   * Developing individual and team action plans

   Supporting self-management skills using:

   Daily interactions • Encouraging problem-solving

   • Enabling use of personal resources

   • Changing focus of therapy

   Patient-held workbook • Peer example 'vignettes'

   • Reflecting on progress

   • Recording aspirations/hopes
   * Small targets

   Adaptions to the Bridges intervention to contextualise to the clinical setting (specialist service) and population (NMDs)
   * Option for remote delivery to mitigate impact of COVID-19
   * Co-production of Bridges resources (workbook/digital tool
   * Health delivery system: intervention optimised for one-off clinical interactions as opposed to multiple rehabilitation sessions
   * Co-design of new educational package for clinicians: Pre-trial consultation with staff at the centre revealed that patients will often only have one or two sessions per year, meaning that the intervention needs to be able to be delivered as part of a one-off session to fit into the structure of the clinical service at Queen Square. Subsequently, the NM Bridges educational package for clinicians (their training in how to deliver the intervention) has been co-designed with key stakeholders so that it can be delivered in a one-off session (rather than in multiple sessions as it has been in previous trials).

ELIGIBILITY:
Inclusion Criteria:

* be over the age of 18
* be a patient at Queen Square Centre for Neuromuscular Diseases or UCLH
* have a diagnosis of Neuromuscular Disease from a neurologist at the Queen Square Centre for Neuromuscular Diseases.
* be those whom their healthcare professionals judge have the capacity to give informed consent to participate in the research.

Exclusion Criteria:

* Patients <18
* Patients that do not attend clinics at Queen Square Centre for Neuromuscular Diseases or UCLH
* Patients that do not have the capacity to provide informed consent
* Patients will be excluded if they have competing comorbidities influencing their rehabilitation, e.g. malignant cancer;
* have significant issues with their readiness to participate as judged by the clinical team, e.g. illness of a carer; did not require multidisciplinary rehabilitation; or had hearing and visual impairments precluding their ability to fully participate in NM Bridges

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview: Feasibility and acceptability of the intervention | Up to 3 months
  Recruitment and participant experience

SECONDARY OUTCOMES:
Euroquol-5D | Up to 3 months
  Quality of life rating scale
Self-Efficacy Scale | Up to 3 months
  Rating scale of confidence and self-efficacy
Nottingham Extended Activities of Daily Living | Up to 3 months
  Rating scale of activity participation
General Health Questionnaire | Up to 3 months
  Rating scale of perception of general health
Oxford Participation and Activities Questionnaire, Ox-PAQ | Up to 3 months
  Rating scale of participation in activities

CONTACTS AND LOCATIONS:
Overall Officials: Gita Ramdharry, Principal Investigator — UCLH NHS Trust
Locations (1):
- Queen Square centre for Neuromuscular Diseases, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No